CLINICAL TRIAL: NCT03944577
Title: Impact of Evolocumab (Repatha) in Cardiac Transplant Patients With Coronary Allograft Vasculopathy
Brief Title: Impact of Evolocumab in Cardiac Transplant Patients With CAV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0104-19-FB
Record Dates: First submitted 2019-04-22; First posted 2019-05-09 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Heart Transplant
Keywords: coronary allograft vasculopathy; lipid; heart transplant; low density lipoprotein; proprotein convertase subtilisin/kexin type 9; PCSK9
MeSH Terms: conditions — Hypercholesterolemia, Autosomal Dominant, 3 | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Evolocumab (Experimental): Patients who will receive the study drug.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Enrolled study participants will be treated with evolocumab (Repatha) 140 mg injected subcutaneously every 2 weeks for 52 weeks. All study participants will receive instruction on correct self-administration by research pharmacists. Study drug will be mailed to patients on a monthly basis for self-administration by patients. The evolocumab dose (140 mg every 2 weeks) will remain constant for the duration of the study. Side effects will be assessed on a quarterly basis. Serious adverse events considered related to treatment, death, and pregnancy will all result in immediate discontinuation of the study drug.
  Other Names: Repatha

SUMMARY:
Coronary allograft vasculopathy (CAV) is diffusely accelerated atherosclerosis of a transplanted heart. Evolocumab (Repatha) is an FDA-approved drug for lowering low density lipoprotein (LDL) in patients who have not received a heart transplant. This drug works as a PCSK9-inhibitor. The primary objective of this study is to measure the impact of PCSK9-inhibitors on serum LDL in heart transplant patients with CAV after 12 weeks compared to baseline.

DETAILED DESCRIPTION:
Heart transplant remains the treatment of choice for patients with advanced heart failure. Coronary allograft vasculopathy (CAV) is diffusely accelerated atherosclerosis of the donor heart, and limits long term survival after transplant. The pathophysiology of CAV is complex and involves smooth muscle proliferation, inflammatory infiltrates, and lipid deposition. To date, only statin therapy has reduced CAV-related mortality. PCSK9 inhibitors are a new lipid lowering therapy shown to reduce cardiovascular clinical events in patients with coronary artery disease. We hypothesize that PCSK9 inhibition via evolocumab will significantly lower low density lipoprotein (LDL) and be well-tolerated in transplant patients with CAV. This phase II, open label, single center trial with enroll up to 40 heart transplant patients with CAV for treatment with evolocumab for one year. The primary outcome will be percent change in LDL at 12 weeks. Secondary outcomes will include change in CAV progression, impact of evolocumab on immunosuppression regimens and transplant rejection, and change in serum lipids after 52 weeks. Results of this study are intended to provide safety data in heart transplant patients with CAV and assess secondary outcomes including CAV progression and impact on immunosuppression and transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients 19-80 years of age
* Coronary allograft vasculopathy grade 1 or 2 documented by left heart cardiac catheterization
* Able to provide signed informed consent

Exclusion Criteria:

* Cardiac allograft vasculopathy (CAV) grade 3
* Rejection requiring IV therapy in the prior 3 months
* Infection requiring IV therapy in the prior 3 months
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal
* Current or recent use of a PCSK9 inhibitor within the past 12 weeks
* Organ transplant recipient other than heart
* Renal dysfunction defined as glomerular filtration rate (GFR) < 20 ml/min
* Known allergy to evolocumab or its components

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Stoller, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available) to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Evolocumab: Heart transplant participant with Cardiac allograft vasculopathy (CAV) who received the study drug.
  Enrolled study participants will be treated with evolocumab (Repatha) 140 mg injected subcutaneously every 2 weeks for 52 weeks.
Period: Overall Study
Arm/Group | Evolocumab
Started | 26
Completed | 23
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- Evolocumab: Heart transplant participants with CAV who received the study drug. Enrolled study participants will be treated with evolocumab (Repatha) 140 mg injected subcutaneously every 2 weeks for 52 weeks.
Arm/Group | Evolocumab
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 63 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Low density lipoprotein (LDL) [Median (Inter-Quartile Range); unit: mg/dL] | 100 [82 to 124]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum LDL (mg/dL) After 12 Weeks of Evolocumab
Description: The primary outcome measure for this study was percent change in LDL from baseline after 12 weeks of evolocumab therapy. Serum LDL was measured at baseline and after 12 weeks of evolocumab therapy. This primary endpoint was used in prior phase 2 trials investigating evolocumab in other patient populations. Wilcoxon matched-pairs signed rank test was used for statistical assessment.
Time Frame: 12 weeks
Population: This single arm study investigated the impact of PCSK9 inhibition via evolocumab on serum LDL in heart transplant patients with CAV after 12 weeks compared to baseline. Percent Change in serum LDL will serve as the primary endpoint for comparison.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Evolocumab: Heart transplant participant with CAV who received the study drug. Enrolled study participants will be treated with evolocumab (Repatha) 140 mg injected subcutaneously every 2 weeks for 52 weeks.
Arm/Group | Evolocumab
Number analyzed (Participants) | 24
percent change | 68 [51 to 82]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were assessed by research personnel at weeks 2, 4, 12, 26, 38 and study conclusion (week 52).
Groups:
- Treatment Arm: Heart transplant participant with CAV who received the study drug. Enrolled study participants will be treated with evolocumab 140 mg injected subcutaneously every 2 weeks for 52 weeks.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 11/26
Other Adverse Events (participants affected / at risk) | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=26)
hospitalization (Infections and infestations) | 3 (3)
hospitalization (Vascular disorders) | 3 (3)
hospitalization (Cardiac disorders) | 3 (3)
hospitalization (Gastrointestinal disorders) | 1 (1)
hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=26)
nausea (Gastrointestinal disorders) | 2
URI/sinus congestion/viral infection (Infections and infestations) | 6
palpitations (Cardiac disorders) | 1
rejection (Cardiac disorders) | 1
myalgia/back pain (Musculoskeletal and connective tissue disorders) | 5
overactive bladder (Renal and urinary disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
phlebitis/urticaria (Skin and subcutaneous tissue disorders) | 2
toothache (Skin and subcutaneous tissue disorders) | 1
headache (Musculoskeletal and connective tissue disorders) | 1
confusion (Nervous system disorders) | 1
fall (Musculoskeletal and connective tissue disorders) | 1
toe fracture (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Cardiac disorders) | 1
hypoglycemia (Endocrine disorders) | 1

LIMITATIONS AND CAVEATS:
The study was a small, single center, one-arm trial. The trial was not randomized or blinded, and did not include a placebo-controlled group due to patient number and financial constraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03944577/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT03944577/ICF_001.pdf